CLINICAL TRIAL: NCT01698398
Title: The Increase Study. Effect of Incremental Versus Fixed Pump on Peak Oxygen Consumption in Heart Failure Patients Supported With a Continuous Flow Left Venticular Assist Device.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Masking: Double
Other Study IDs: H-1-2012-092
Record Dates: First submitted 2012-10-02; First posted 2012-10-03 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2012-10

CONDITIONS: Heart Failure.
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- CF-LVAD pumpspeed. (Experimental): Optimal pumpspeed setting of CF-LVAD during exercise on ergometric bicycle.
  Interventions: Device: Incremental pump speed of CF-LVAD.

INTERVENTIONS:
Device: Incremental pump speed of CF-LVAD. — Peak oxygen consumption with fixed versus incremental pump speed.
  Other Names: HeartMate II.

SUMMARY:
The purpose of the study is to examine the relationship between working capacity (peak oxygen consumption) and pump speed of continuous flow left ventricular assist devices (CF-LVADs)in heart failure patients. The hypothesis is that it is possible to increase peak oxygen consumption by incrementally increasing CF-LVAD pumpspeed during exercise.

The study population will consist of severe heart failure patients with CF-LVADs treated at The Heart Centre of Copenhagen University Hospital Rigshospitalet.

ELIGIBILITY:
Inclusion Criteria:

* HeartMate II patients who underwent surgery and follow-up at The Heart Centre of Rigshospitalet.
* Heart failure in stable phase without the need for intravenous inotropic therapy.
* Ischemic and non-ischemic cardiomyopathy.

Exclusion Criteria:

* Severe aortic insufficiency.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2012-10; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Peak oxygen consumption. | Day 1
  ml oxygen/minute/kg

SECONDARY OUTCOMES:
Working capacity. | Day 1
  Watt

OTHER OUTCOMES:
Exercise time (minutes), anerobic threshold. | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Copenhagen University Hospital, Rigshospitalet., Copenhagen, Denmark

REFERENCES:
- [Derived] Jung MH, Hansen PB, Sander K, Olsen PS, Rossing K, Boesgaard S, Russell SD, Gustafsson F. Effect of increasing pump speed during exercise on peak oxygen uptake in heart failure patients supported with a continuous-flow left ventricular assist device. A double-blind randomized study. Eur J Heart Fail. 2014 Apr;16(4):403-8. doi: 10.1002/ejhf.52. PMID 24464845